CLINICAL TRIAL: NCT05022277
Title: Empowering Girls: Health-seeking Behavior, Staying in School and Preventing Risky Sex
Brief Title: Empowering Girls: Health-seeking Behavior, Staying in School, and Preventing Risky Sex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Young 1ove (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Y1HPDME2021
Record Dates: First submitted 2021-08-11; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy Related; Behavior, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phone-based intervention Plus SMS messages (Experimental)
  Interventions: Behavioral: Low tech health Phone + SMS messages
- SMS messages only (Experimental)
  Interventions: Behavioral: Low tech health SMS messages
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Low tech health SMS messages — Weekly health-related SMS messages are provided to adolescents.
  Arms: SMS messages only
Behavioral: Low tech health Phone + SMS messages — Weekly health-related phone calls plus SMS messages are provided to adolescents.
  Arms: Phone-based intervention Plus SMS messages

SUMMARY:
This study will test the effectiveness of a phone-based big sister/big brother program designed to provide health information and support, reduce school dropouts, and promote safer relationships.

The program's goal is to create a phone-based safe space, to ensure adolescents remained connected with access to support and health information during COVID lockdowns.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent who provided their phone number to Young 1ove staff when prompted by their school; or their siblings/ other adolescents living in the same household.
* Parents and students consented to participate.

Exclusion Criteria:

-

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Share of students that have been or are pregnant and/or have dropped out of school | ~6 months post-program
  These two outcomes (using school administrative data on whether students have dropped out of school and were pregnant) will be combined into a composite variable equal to 1 if the student has become pregnant and/or has dropped out of school.
Share of students with the accurate belief that older partners have the highest risk of HIV compared to younger partners. | ~4 weeks post program
  Indicator variable from the survey question wording: "Who do you think has the highest risk of infecting you with HIV?"

SECONDARY OUTCOMES:
Share of students reporting that they make the final decision in their life about visiting a Sexual and reproductive health clinic | ~4 weeks post program
  Indicator variable from the survey question response
Share of students reporting that if they or their partner were pregnant, they would tell the data collector | ~4 weeks post program
  Indicator variable coded 1 if student answered likely or very likely to 'If you were pregnant, how likely would you be to tell me?'

OTHER OUTCOMES:
Share of students disclosing personal information to the data collector in the open-ended question at the end of the survey. | ~4 weeks post program
Share of female students reporting that they agree or strongly agree with the statement 'If I don't want to hold hands with a guy, I can comfortably refuse to do it' | ~4 weeks post program
Share of students listing known support services when asked 'If a friend experienced dating difficulties or violence, do you know any organizations, services or phone numbers you could suggest she contact to get some help if she wanted?' | ~4 weeks post program

CONTACTS AND LOCATIONS:
Overall Officials: Noam Angrist, PhD, Study Chair — University of Oxford
Locations (1):
- Young 1ove, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No